CLINICAL TRIAL: NCT01422720
Title: Safety and Efficacy of Eslicarbazepine Acetate (ESL) as Adjunctive Therapy for Partial Seizures in Elderly Patients
Brief Title: Safety and Efficacy of Eslicarbazepine Acetate as Adjunctive Therapy for Partial Seizures in Elderly Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-401; 0140BI17.MPB (Other: SCOPE); 2009-012587-14 (EudraCT Number)
Record Dates: First submitted 2011-07-29; First posted 2011-08-24 (Estimated); Results first posted 2014-07-18 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-06

CONDITIONS: Epilepsy
Keywords: Epilepsy; ESL; Eslicarbazepine Acetate; BIAL; BIA; Partial-onset Seizures
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eslicarbazepine Acetate tablets (800 mg) (Experimental)
  Interventions: Drug: Eslicarbazepine Acetate

INTERVENTIONS:
Drug: Eslicarbazepine Acetate — ESL tablets (800 mg) QD
  Other Names: Zebinix

SUMMARY:
This is an open Label study to investigate the safety and efficacy of eslicarbazepine acetate as adjunctive therapy for partial seizures in elderly patients.

DETAILED DESCRIPTION:
Multicenter study in approximately 100 elderly patients. The study will follow an open-label design and will consist of 8-week baseline period, followed by a 26-week treatment period and a 4-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent form;
2. Of age 65 years or older;
3. A documented diagnosis of epilepsy for at least 12 months,
4. At least 2 partial-onset seizures (including subtypes of simple partial, complex partial and/or partial seizures evolving to secondarily generalised) in the 4 weeks prior to screening;
5. Currently treated with 1 or 2 AEDs (any except oxcarbazepine) in a stable dosage regimen for at least 4 weeks prior to screening. Vagus nerve stimulation (VNS) is to be considered as an AED (i.e., only one concomitant AED is allowed in patients with VNS);
6. Willing and able to comply with all trial requirements, in the judgment of the investigator;
7. At least 2 partial-onset seizures (documented in the diary) per 4 weeks during the 8-week baseline period;
8. Satisfactorily complied with the study requirements during the baseline period

Exclusion Criteria:

1. Only simple partial seizures with no motor symptomatology (classified as A2-4) according to the International Classification of Epileptic Seizures);
2. Primarily generalised seizures;
3. Known progressive neurological disorders (progressive brain disease, epilepsy secondary to progressive central nervous system lesion) and progressive dementia;
4. Occurrence of seizures too close to count accurately;
5. History of status epileptic or cluster seizures 8i.e. 3 or more seizures within 30 minutes) within the 3 months prior to screening;
6. Seizures of non-epileptic origin;
7. Major psychiatric disorders;
8. History of suicide attempt;
9. Currently treated with oxcarbazepine;
10. Previous use of ESL or participation in a clinical study with ESL;
11. Known hypersensitivity to other carboxamide derivatives (e.g. oxcarbazepine, carbamazepine) or to any of the excipients;
12. Uncontrolled cardiac, renal, hepatic, endocrine, gastrointestinal, metabolic, haematological or oncology disorder, hypo - or hyper thyroidism of any type;
13. Second or third-degree atrioventricular blockade or any clinically significant abnormality in the 12-lead electrocardiogram (ECG) as determined by the investigator;
14. Relevant clinical laboratory abnormalities as determined by the investigator (e.g. plasma sodium <130 mmol/L, alanine or aspartate aminotransferases >2.0 times above the upper limit of the range, or white blood cell count <3,000 cells/mm3;
15. Calculated creatinine values < 30 mL/min at screening;
16. Any other condition or circumstance that, in the opinion of the investigator, may compromise the patient's ability to comply with the study protocol;
17. Received an investigational drug (or a medical device) within 3 months of screening or is currently participating in another trial of an investigational drug (or medical device) trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- Austria (3):
  - Universitätsklinik für Neurologie; Arbeitsgruppe Epileptologie, Innsbruck
  - Universitätsklinik für Neurologie; Christian-Doppler-Klinik, Salzburg
  - Medizinische Universitat Wien Klinik fur Neurologie, Vienna
- Bulgaria (6):
  - 4 MHAT Sofia, Sofia
  - Diagnostic & Consultative Center "Sveta Anna" EOOD, Sofia
  - First MHAT-Sofia, Sofia
  - UMHAT "Aleksandrovska", Sofia
  - UMHAT "Tsaritsa Yoanna -ISUL", Sofia
  - MHAT "Prof. Stoyan Kirkovich", Stara Zagora
- Croatia (3):
  - General County Hospital Požega, Neurology department, Požega
  - Polyclinic for neurology and psychiatry 'Interneuron, Rijeka
  - Clinical Hospital Centre Split, Split
- Czechia (7):
  - Neurologická klinika, FN u Sv. Anny, Brno
  - NZZ BORMED s.r.o., Ostrava - Třebovice
  - Neurologická ambulance, Pilsen
  - Clintrial, s.r.o., Prague
  - Medical Services Prague s.r.o., Prague
  - Oddělení neurologie, FN Bulovka, Prague
  - Fakultní Thomayerova nemocnice s poliklinikou, Neurologická klinika, Praha 4 - Krč
- France (3):
  - Hôpital Gui de Chauliac, Explorations neurologiques et d'épileptologie, Montpellier
  - Hôpital Central - Service de Neurologie, Nancy
  - Groupement Hospitalier Universitaire Est, Pitié-Salpétrière; Clinique des Maladies du Système Nerveux, Paris
- Germany (7):
  - Klinik für Epileptologie Universität Bonn, Bonn
  - Zentrum Epilepsie Erlangen, Erlangen
  - Diakonie Kork, Epilepsiezentrum, Kehl-Kork
  - IZKS; Universitätsmedizin der Johannes-Gutenberg-Universität Mainz, Mainz
  - Studienzentrum Dr. Stephan Arnold, München
  - Neurologische Gemeinschaftspraxis am Seelberg, Stuttgart
  - Universitäts- und Rehabilitationskliniken Ulm (RKU), Klinik für Neurologie, Ulm
- Poland (4):
  - "Klinika Neurologii Rozwojowej, Gdansk
  - Centrum Leczenia Padaczki i Migreny, Krakow
  - Małopolskie Centrum Medyczne s.c., Krakow
  - Centrum Terapii Współczesnej, Lodz
- Portugal (5):
  - AIBILI - Centro de Estudos de Biodisponibildade, Coimbra
  - Centro Hospitalar de Lisboa Norte, EPE - Hospital de Staª Maria - Centro de Estudos Egas Moniz, Lisbon
  - Centro Hospitalar de Lisboa Ocidental, EPE - Hospital Egas Moniz, Lisbon
  - Unidade Local de Saúde de Alto Minho, EPE - Hospital de Santa Luzia - Serviço de Neurologi, Viana do Castelo
  - Centro Hospitalar de Trás-os -Montes e Alto-Douro, EPE - Hospital de São Pedro - Serviço de Neurologia, Vila Real
- Romania (4):
  - C.M.D.T.A. Neomed, Brasov
  - Cabinet Medical Individual "Dr. Roceanu Adina Maria" -Neurologie, Neurofiziologie (EEG, EMG, PEC), Bucharest
  - Sc Clubul Sanatatii Srl, Campulung Muscel
  - Spitalul Clinic de Neuropsihiatrie Craiova, Craiova; Jud. Dolj
- Spain (6):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - IMAS Hospital del Mar, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Virgen Macarena, Seville

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 44 clinical centres in Europe and Asia.
  Studied period (years):
  Date of first enrolment: 19-APR-2010 Date of last subject completed: 08-OCT-2013
Pre-assignment Details: In this trial all subjects received the same treatment.
Groups:
- Esl 800 mg: Eslicarbazepine Acetate (Esl) tablets (800 mg) QD
Period: Overall Study
Arm/Group | Esl 800 mg
Started | 72
Safety Set | 72
Full Analysis Set (FAS) | 71
Per-Protocol Set (PPS) | 55
Completed | 50
Not Completed | 22
Not completed — Adverse Event | 16
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 4
Not completed — Ineligibility | 1

BASELINE CHARACTERISTICS:
Arm/Group | Esl 800 mg
Number analyzed (Participants) | 72
Age, Customized [Number; unit: participants]
  65-69 years | 30
  70-74 years | 19
  75-79 years | 19
  80-84 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Reported Adverse Events (AE)
Description: An AE was defined as Treatment-Emergent Adverse Event (TEAE), if first onset or worsening was after the first intake of investigational medicinal product (IMP) and not more than 14 days after the last administration of IMP.
  TEAE assessment:
  * patients who died
  * patients who died due to Treatment-emergent adverse event (TEAE)
  * patients with at least one Serious Adverse Event (SAE)
  * patients with at least one Treatment-emergent Serious Adverse Event (TESAE)
  * patients prematurely terminated due to TEAE
  * patients with at least one TEAE
  * patients with at least one related TEAE
  * patients with at least one severe TEAE
  * patients without any TEAE
Time Frame: throughout the study
Measure: Number; unit: participants
Arm/Group | Esl 800 mg
Number analyzed (Participants) | 72
participants
  patients who died | 3
  patients who died due to TEAE | 3
  patients with at least one SAE | 11
  patients with at least one TESAE | 10
  patients prematurely terminated due to TEAE | 18
  patients with at least one TEAE | 47
  patients with at least one related TEAE | 31
  patients without any TEAE | 25
  patients with at least one severe TEAE | 12

2. Secondary Outcome: Change From Baseline in Standardized Seizure Frequency
Description: Absolute and relative changes from baseline of seizure frequency standardised to a frequency per 4 weeks.
Time Frame: 8-week Baseline Period and 26-week Treatment Period
Measure: Mean (Standard Deviation); unit: seizures/4 weeks
Groups:
- FAS - Baseline Period; FAS - Treatment Period: The Full Analysis Set (FAS) consisted of all subjects who received at least one dose of IMP and had at least one day of seizure evaluation reported in the patient diary after Visit 2.
- PPS - Baseline Period; PPS- Treatment Period: The Per Protocol Set (PPS) consisted of all subjects in the FAS who had completed the Treatment Period and did not have any protocol deviation (e.g. poor compliance, diaries not properly filled) in a sufficiently serious manner to warrant data (but not subject) exclusion.
Arm/Group | FAS - Baseline Period | FAS - Treatment Period | PPS - Baseline Period | PPS- Treatment Period
Number analyzed (Participants) | 71 | 71 | 55 | 55
seizures/4 weeks | 4.8 (5.53) | 3.6 (5.84) | 4.0 (3.54) | 3.1 (5.64)

ADVERSE EVENTS:
Time Frame: Throughout the study
Arm/Group | Esl 800 mg
Serious Adverse Events (participants affected / at risk) | 11/72
Other Adverse Events (participants affected / at risk) | 43/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esl 800 mg (N=72)
Altered state of consciousness (Nervous system disorders) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Postictal psychosis (Psychiatric disorders) | 1 (1)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esl 800 mg (N=72)
Dizziness (Nervous system disorders) | 9 (11)
Somnolence (Nervous system disorders) | 7 (7)
Fatigue (General disorders) | 6 (7)
Convulsion (Nervous system disorders) | 6 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (6)
Nasopharyngitis (Infections and infestations) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other